CLINICAL TRIAL: NCT03528954
Title: Effectivity of 0.5 mg/kg Propofol in the End of Anesthesia to Reduce the Incidence of Postanesthetic Emergence Agitation in Pediatric Patients Under General Inhalation Anesthesia
Brief Title: Propofol to Reduce the Incidence of Postanesthetic Emergence Agitation in Pediatric Patients Under General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Andi Ade Wijaya Ramlan, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes022
Record Dates: First submitted 2018-04-27; First posted 2018-05-18 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Pediatric ALL
Keywords: Emergence agitation; Propofol; General anesthesia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Emergence Delirium | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol (Active Comparator): Received intravenous 0.5mg/kg propofol
  Interventions: Drug: Propofol
- Control (No Intervention): Do not received intravenous 0.5 mg/kg propofol

INTERVENTIONS:
Drug: Propofol — Those who received intravenous propofol
  Arms: Propofol

SUMMARY:
This study aimed to know the effectivity of 0.5 mg/kg propofol in the end of anesthesia to reduce the incidence of postanesthetic emergence agitation in pediatric patients under general inhalation anesthesia

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine Universitas Indonesia was acquired prior conducting the study. Subjects were given informed consent before enrolling the study and randomized into two groups; propofol and control. Non-invasive blood pressure monitor, electrocardiogram (ECG), pulse-oxymetry, and capnograph were set on the subjects in the operation room. Induction and maintenance of anesthesia will use sevoflurane. Mechanical ventilation will be given to maintaining end-tidal carbon dioxide 35 to 40 mmHg. After surgery, patient will be given intravenously 15mg/kg acetaminophen, 0.05mg/kg neostigmine, and 0.02 mg/kg atropine. Patient will also be given propofol 0.5 mg/kg on propofol group while no propofol will be given on control group. 30 minutes after patient was admitted to post-anesthesia care unit, patient will be evaluated for emergence agitation using Aono scale and Pediatric Anesthesia Emergence Delirium scale. The incidence of emergence agitation, hypotension, and desaturation will be treated accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing non-emergency surgery with general anesthesia
* Patient using sevoflurane as anesthetic agent
* Patient aged 1 - 5 years old
* American Society of Anesthesiologists (ASA) physical status 1 - 2
* Patient family signed the informed consent to be included in the study

Exclusion Criteria:

* Patient that will undergo ophthalmologic and otorhinolaryngologic surgery
* Patient that will require post operation stay in Intensive Care Unit
* Patient with psychological and neurological problem
* Patient with developmental delay
* Patient using sedative drugs
* Patient with allergy to propofol
* Patient or patient family with history of malignant hyperthermia
* Patient with difficulty on intubation and ventilation
* Patient with cardiovascular disease
* Patient with hemodynamic instability

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence of emergence agitation | 30 minutes after being admitted to post anesthesia care unit
  Evaluated using Aono scale and Pediatric Anesthesia Emergence Delirium (PAED) scale. Patients with ≥3 on Aono scale AND ≥10 on PAED scale are diagnosed as emergence agitation

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Hoff SL, O'Neill ES, Cohen LC, Collins BA. Does a prophylactic dose of propofol reduce emergence agitation in children receiving anesthesia? A systematic review and meta-analysis. Paediatr Anaesth. 2015 Jul;25(7):668-76. doi: 10.1111/pan.12669. Epub 2015 Apr 27. PMID 25917689
- [Background] Costi D, Ellwood J, Wallace A, Ahmed S, Waring L, Cyna A. Transition to propofol after sevoflurane anesthesia to prevent emergence agitation: a randomized controlled trial. Paediatr Anaesth. 2015 May;25(5):517-23. doi: 10.1111/pan.12617. Epub 2015 Jan 13. PMID 25586124
- [Background] Jiang S, Liu J, Li M, Ji W, Liang J. The efficacy of propofol on emergence agitation--a meta-analysis of randomized controlled trials. Acta Anaesthesiol Scand. 2015 Nov;59(10):1232-45. doi: 10.1111/aas.12586. Epub 2015 Aug 6. PMID 26251008
- [Background] Aouad MT, Yazbeck-Karam VG, Nasr VG, El-Khatib MF, Kanazi GE, Bleik JH. A single dose of propofol at the end of surgery for the prevention of emergence agitation in children undergoing strabismus surgery during sevoflurane anesthesia. Anesthesiology. 2007 Nov;107(5):733-8. doi: 10.1097/01.anes.0000287009.46896.a7. PMID 18073548
- [Background] Dahmani S, Stany I, Brasher C, Lejeune C, Bruneau B, Wood C, Nivoche Y, Constant I, Murat I. Pharmacological prevention of sevoflurane- and desflurane-related emergence agitation in children: a meta-analysis of published studies. Br J Anaesth. 2010 Feb;104(2):216-23. doi: 10.1093/bja/aep376. Epub 2010 Jan 3. PMID 20047899
- [Background] Huett C, Baehner T, Erdfelder F, Hoehne C, Bode C, Hoeft A, Ellerkmann RK. Prevention and Therapy of Pediatric Emergence Delirium: A National Survey. Paediatr Drugs. 2017 Apr;19(2):147-153. doi: 10.1007/s40272-017-0212-x. PMID 28130755
- [Background] Kanaya A, Kuratani N, Satoh D, Kurosawa S. Lower incidence of emergence agitation in children after propofol anesthesia compared with sevoflurane: a meta-analysis of randomized controlled trials. J Anesth. 2014 Feb;28(1):4-11. doi: 10.1007/s00540-013-1656-y. Epub 2013 Jun 26. PMID 23800983
- [Background] Moore AD, Anghelescu DL. Emergence Delirium in Pediatric Anesthesia. Paediatr Drugs. 2017 Feb;19(1):11-20. doi: 10.1007/s40272-016-0201-5. PMID 27798810
- [Background] Kanaya A. Emergence agitation in children: risk factors, prevention, and treatment. J Anesth. 2016 Apr;30(2):261-7. doi: 10.1007/s00540-015-2098-5. Epub 2015 Nov 24. PMID 26601849
- [Background] Chidambaran V, Costandi A, D'Mello A. Propofol: a review of its role in pediatric anesthesia and sedation. CNS Drugs. 2015 Jul;29(7):543-63. doi: 10.1007/s40263-015-0259-6. PMID 26290263
- [Background] Ali MA, Abdellatif AA. Prevention of sevoflurane related emergence agitation in children undergoing adenotonsillectomy: A comparison of dexmedetomidine and propofol. Saudi J Anaesth. 2013 Jul;7(3):296-300. doi: 10.4103/1658-354X.115363. PMID 24015133
- [Background] Makkar JK, Bhatia N, Bala I, Dwivedi D, Singh PM. A comparison of single dose dexmedetomidine with propofol for the prevention of emergence delirium after desflurane anaesthesia in children. Anaesthesia. 2016 Jan;71(1):50-7. doi: 10.1111/anae.13230. Epub 2015 Oct 7. PMID 26444149
- [Background] Silva LM, Braz LG, Modolo NS. Emergence agitation in pediatric anesthesia: current features. J Pediatr (Rio J). 2008 Mar-Apr;84(2):107-13. doi: 10.2223/JPED.1763. PMID 18372935
- [Background] Smith HA, Fuchs DC, Pandharipande PP, Barr FE, Ely EW. Delirium: an emerging frontier in the management of critically ill children. Anesthesiol Clin. 2011 Dec;29(4):729-50. doi: 10.1016/j.anclin.2011.09.011. PMID 22078920
- [Background] Maldonado JR. Neuropathogenesis of delirium: review of current etiologic theories and common pathways. Am J Geriatr Psychiatry. 2013 Dec;21(12):1190-222. doi: 10.1016/j.jagp.2013.09.005. PMID 24206937
- [Background] Aono J, Mamiya K, Manabe M. Preoperative anxiety is associated with a high incidence of problematic behavior on emergence after halothane anesthesia in boys. Acta Anaesthesiol Scand. 1999 May;43(5):542-4. doi: 10.1034/j.1399-6576.1999.430509.x. PMID 10342002
- [Background] Beringer RM, Greenwood R, Kilpatrick N. Development and validation of the Pediatric Anesthesia Behavior score--an objective measure of behavior during induction of anesthesia. Paediatr Anaesth. 2014 Feb;24(2):196-200. doi: 10.1111/pan.12259. Epub 2013 Sep 19. PMID 24103068
- [Background] Burke CN, Voepel-Lewis T, Hadden S, DeGrandis M, Skotcher S, D'Agostino R, Walton S, Malviya S. Parental presence on emergence: effect on postanesthesia agitation and parent satisfaction. J Perianesth Nurs. 2009 Aug;24(4):216-21. doi: 10.1016/j.jopan.2009.03.014. PMID 19647657
- [Background] Singh R, Kharbanda M, Sood N, Mahajan V, Chatterji C. Comparative evaluation of incidence of emergence agitation and post-operative recovery profile in paediatric patients after isoflurane, sevoflurane and desflurane anaesthesia. Indian J Anaesth. 2012 Mar;56(2):156-61. doi: 10.4103/0019-5049.96325. PMID 22701207
- [Background] Voepel-Lewis T, Malviya S, Tait AR. A prospective cohort study of emergence agitation in the pediatric postanesthesia care unit. Anesth Analg. 2003 Jun;96(6):1625-1630. doi: 10.1213/01.ANE.0000062522.21048.61. PMID 12760985
- [Background] Key KL, Rich C, DeCristofaro C, Collins S. Use of propofol and emergence agitation in children: a literature review. AANA J. 2010 Dec;78(6):468-73. PMID 21309294
- [Background] Sikich N, Lerman J. Development and psychometric evaluation of the pediatric anesthesia emergence delirium scale. Anesthesiology. 2004 May;100(5):1138-45. doi: 10.1097/00000542-200405000-00015. PMID 15114210
- [Background] Kim MS, Moon BE, Kim H, Lee JR. Comparison of propofol and fentanyl administered at the end of anaesthesia for prevention of emergence agitation after sevoflurane anaesthesia in children. Br J Anaesth. 2013 Feb;110(2):274-80. doi: 10.1093/bja/aes382. Epub 2012 Oct 26. PMID 23103775
- [Background] Liu GY, Chen ZQ, Zhang ZW. Comparative study of emergence agitation between isoflurane and propofol anesthesia in adults after closed reduction of distal radius fracture. Genet Mol Res. 2014 Jan 24;13(4):9285-91. doi: 10.4238/2014.January.24.9. PMID 24615079